CLINICAL TRIAL: NCT02035449
Title: Video Laryngoscopy in Pre-hospital Critical Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: McGrath MAC 1
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-12

CONDITIONS: Airway Morbidity; Airway Disease; Respiratory Insufficiency; Respiratory Failure
Keywords: Video laryngoscope; Pre-hospital; Endotracheal intubation; Difficult endotracheal intubation; Pre hospital Critical care; McGrath MAC; Airway device
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- McGrath MAC: McGrath MAC is a videolaryngscope
  Interventions: Device: McGrath MAC

INTERVENTIONS:
Device: McGrath MAC — McGrath MAC is a videolaryngoscope

SUMMARY:
Difficult conditions and critically ill and injured patients may complicate endotracheal intubation in the pre-hospital setting. The incidence of complications increase when two or more endotracheal intubation attempts are needed.

The aim of this study is to estimate the incidence of difficult pre-hospital endotracheal intubation after the introduction of the McGrath MAC Video laryngoscope as the primary airway device for pre-hospital endotracheal intubation.

Hypothesis:

• In our pre-hospital critical care teams, staffed with experienced anaesthesiologists, the rate of difficult PHETI (defined as more than one intubation attempt needed to secure a patent airway) is lower than 10 %, when using the McGrath MAC VL as primary choice in pre-hospital intubations.

ELIGIBILITY:
Inclusion Criteria:

* Patients where the anaesthesiologists on the participating pre-hospital critical care teams attempt prehospital endotracheal intubation.

Exclusion Criteria:

* Patients< 15 years of age

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the Central Region of Denmark where the anaesthesiologists on the participating pre-hospital critical care teams attempt prehospital endotracheal intubation.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of difficult pre-hospital endotracheal intubation | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mads P Vandborg, Doctor, Principal Investigator — Pre-hospital Medical Services, Central Denmark Region
Locations (1):
- Pre-hospital Medical Services, Central Denmark Region, Aarhus, Denmark